CLINICAL TRIAL: NCT06653335
Title: EFFECTIVENESS of the EDUCATION SUPPORT PROGRAM VIA TEXT MESSAGE
Brief Title: Effectiveness of the Education Support Program Provided Via Text Message
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MarmaraUEBE2
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Midwifery Students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): All students to be included in the study will be pre-tested through Google Form's. After the pre-test, the students in the experimental group will be sent images created by the researchers via text message for 4 weeks (22 days) and consisting of the information given in the Basic Principles and Practices in Midwifery Course. Each visual will contain one piece of information. The researchers will send 6 visuals to the students in the experimental group via text message every day for 4 weeks, except Saturdays and Sundays. The post-test will be applied immediately after the end of the implementation process. The messages will be short and contain a single piece of information.
  Interventions: Behavioral: Education Support Programme via Text Message
- Control Group (No Intervention): No treatment will be carried out.

INTERVENTIONS:
Behavioral: Education Support Programme via Text Message — All students to be included in the study will be pre-tested via Google Form's. After the pre-test, the students in the experimental group will be sent images created by the researchers via text message for 4 weeks (22 days) and consisting of the information given in the Basic Principles and Practices in Midwifery Course. Each visual will contain one piece of information. The researchers will send 6 visuals to the students in the experimental group via text message every day for 4 weeks, except Saturdays and Sundays. The post-test will be applied immediately after the end of the implementation process. The messages will be short and contain a single piece of information.
  Arms: Experimental Group

SUMMARY:
Information will be provided to first year midwifery students via text message within the scope of the 'Basic Principles and Practice in Midwifery Education' support programme. This information is planned to last approximately 4 weeks. The study will be conducted to evaluate the effect of the information provided on the knowledge levels of the students.

ELIGIBILITY:
Inclusion Criteria:

* In 2023-2024 Spring Term, with the success of the Basic Principles and Practices Course in Midwifery to have completed the programme,
* Having a mobile phone,
* Accepting to participate in the research is one of the inclusion criteria of this studyc

Exclusion Criteria:

* Students who incompletely completed the post-test and first test scales will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge Measurement Questionnaire | Before and immediately after education
  The knowledge measurement questionnaire prepared by the researchers according to the curriculum of the related course consists of 133 questions in total. There are 'Yes' or 'No' choices in the questions. Out of 33 questions, those who give the correct answer will be scored as 1 and those who give the wrong answer will be scored as 0. The knowledge measurement questionnaire will be applied in pre-test and post-test. The pre-test will be applied just before the start of the study and the post-test will be applied just after the end of the implementation process.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang, C. S. J., Yang, S. J. H., Chiang, T. H. C., & Su, A. Y. S. (2016). Effects of Situated Mobile Learning Approach on Learning Motivation and Performance of EFL Students. Educational Technology & Society, (2016), 19 (1), 263-276.)
- [Background] Hardini, M. G., Khaizure, T., & Godwin, G. (2024). Exploring the Effectiveness of E-Learning in Fostering Innovation and Creative Entrepreneurship in Higher Education. Startupreneur Business Digital (SABDA Journal), 3(1), 34-42. https://doi.org/10.33050/sabda.v3i1.441
- [Background] Kavruk Y. (2018). Uzaktan Öğrenenlerin Kısa Mesaj ile Eğitsel Destek Sağlanmasına Yönelik Memnuniyetleri ve Öğrenme Düzeyleri. Anadolu Üniversitesi Sosyal Bilimler Enstitüsü, Yüksek Lisans Tezi. Eskişehir. 2018.